CLINICAL TRIAL: NCT00341081
Title: Validation of Self-Reported Needle Sharing Among Injection Drug Users
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903029; 03-C-N029
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Viral Infection
Keywords: Short Tandem Repeat; Molecular Epidemiology; Viral Infection; Mixture Detection; Intervention & Education; Intervention; Education
MeSH Terms: conditions — Virus Diseases

SUMMARY:
This study, conducted at the Johns Hopkins University School of Public Health in Baltimore, Maryland, will determine how accurately injection drug users report their needle-sharing behavior. Needle-sharing is a major cause of blood-borne diseases, including HIV and hepatitis. Therefore, a better understanding of this behavior is critical for devising strategies to reduce disease spread in this way. Research on needle-sharing behavior has relied heavily on users' self-reports. This study will compare these self-reports with results of DNA tests that show whether a needle has been used by one or more individuals.

Injection drug users 18 years of age or older participating in the Baltimore Needle Exchange Program (BNEP) have been recruited for this study. Syringes distributed to users through the BNEP are collected after use and tested to differentiate between single versus multiple users. The findings are compared with the participants' responses about whether or not they shared their needles and syringes.

Participants visit the clinic every 6 months for an interview, including questions about their mental and physical health, drug use, sexual activity and knowledge about HIV (the virus that causes AIDS) and AIDS. After the interview, a small amount of blood is drawn for testing for HIV, hepatitis, syphilis and other infectious diseases. Some of the blood is stored for future testing. Participants return to the clinic 4 weeks after the interview and blood drawing to get their test results. At this time, they are offered referral for drug treatment, free condoms, advice about drug use and safer sex and an opportunity to ask questions about their health. Participation in the study may continue for up to 5 years.

DETAILED DESCRIPTION:
Needle sharing is a major cause of blood-borne diseases making understanding needle sharing behavior imperative to devising strategies to reduce the disease burden. A DNA-based method, using highly informative genetic markers of short tandem repeats (STRs) is being proposed as a gold standard measure to identify single-use and multi-use syringes. Self-reports of needle sharing, which have been the main source of sharing information for research, will be compared to the genotypic results to validate the responses on such risk behavior. Genotypic information from four autosomal STRs will be used to differentiate DNA from a single versus multiple individuals in syringe exudates obtained from injection drug users (IDUs) from the Baltimore needle exchange program (BNEP) studied by ALIVE II. Detecting three or more distinct alleles at an autosomal STR in the syringe exudates provides evidence that the syringe has been shared by at least two individuals. Matching probabilities will be used to match the genotypic profile of the individual(s) checking in and returning the syringe to allele(s) observed in the syringe exudates, and a mixture discrimination probability will be used to measure the likelihood of single vs. multi genome in the syringe samples. Behavioral surveillance to document the rapid spread of infectious disease from needle sharing among high-risk sub-population such as IDUs are critical for global public health along with the development and implementation of timely interventions.

ELIGIBILITY:
* INCLUSION CRITERIA:

All efforts in BNEP and ALIVE were made to recruit as many IDUs as possible without any discrimination based on sex or race.

EXCLUSION CRITERIA:

Individuals under 18 years of age have been excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442
Dates: Start 2002-10; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Background] Rezza G, Pizzuti R, De Campora E, De Masi S, Vlahov D. Tetanus and injections drug use: rediscovery of a neglected problem? Eur J Epidemiol. 1996 Dec;12(6):655-6. doi: 10.1007/BF00499469. No abstract available. PMID 8982630